CLINICAL TRIAL: NCT05701410
Title: Prevalence of Cardiac Amyloidosis Among Patients With a History of Lumbar Spinal Stenosis.
Acronym: CASS-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steen Hvitfeldt Poulsen (Other)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, Professor, PhD, DMSci, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1-10-72-117-22
Record Dates: First submitted 2023-01-16; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Amyloidosis; Spinal Stenosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Spinal Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients with a history of lumbar spinal stenosis.
  Interventions: Diagnostic Test: DPD scintigraphy

INTERVENTIONS:
Diagnostic Test: DPD scintigraphy — Bone tracer scintigraphy, diagnostic for transthyretin amyloidosis.

SUMMARY:
The study investigates the prevalence of cardiac amyloidosis among patients with a history of lumbar spinal stenosis within the last ten years in the region of central Denmark.

ELIGIBILITY:
Inclusion Criteria:

* History of lumbar spinal stenosis.
* Age > 60 years at the time of spinal stenosis surgery.
* Written informed consent.

Exclusion Criteria:

* Known amyloidosis
* Myelomatosis
* Monoclonal gammopathy of unknown origin, MGUS
* Morbus Waldenstrøm

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of cardiac amyloidosis | 1 year
  DPD scintigraphy with a Perugini Grade 2 og higher.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No